CLINICAL TRIAL: NCT04344301
Title: The Impact of Sharing Audio Recorded Clinic Visits on Self-management in Older Adults: a Multi-site Trial
Brief Title: The Impact of Sharing Audio Recorded Clinic Visits on Self-management in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: The University of Texas Medical Branch, Galveston (Other); Vanderbilt University Medical Center (Other); Dartmouth College (Other); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Paul J. Barr, Assistant Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D20072; 1R56AG061522-01A1 (NIH)
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: Audio recording; Diabetes Mellitus; Hypertension; Patient-centered communication; Self-management; Older adults
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — Sound Recordings

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to AUDIO or UC alone using a block-randomization technique with the clinician acting as the blocking variable; this strategy will ensure an equal number of patients per clinician will be randomly assigned to each study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AUDIO (Experimental): Participant clinic visits will be audio recorded locally on a secure, HIPAA-compliant server. Patient access to recordings will be performed via a secure web-based platform.
  Additionally, participants will be offered the After Visit Summary (AVS) prior to clinic departure, per Usual Care (UC)
  Interventions: Other: Audio recording
- Usual Care (No Intervention): During the trial, patients will be offered to receive the AVS prior to clinic departure as is the current standard at each site.

INTERVENTIONS:
Other: Audio recording — The investigators will audio record the visits of patients in the intervention group. An RA will enter the exam room and begin the recording with the patient's permission. The patient and clinician can choose to stop or start the recording at any time. Once the visit is complete, the RA will enter the room, turn off the recording, and bring the patient to a private room where the RA will follow standardized instructions demonstrating how to access recordings. Patient access to recordings will be possible via a secure web-based platform. Patients will also receive reminders to listen to their recordings.
  Arms: AUDIO

SUMMARY:
The investigators will conduct a multi-site, two-arm, parallel-group, patient-randomized, blocked, controlled, pilot trial with a 3-month follow up in older adults (≥65 years) with diabetes and hypertension. Participants will be randomized to receive AUDIO recordings of their clinic visits (AUDIO) in addition to After Visit Summary (AVS), or their AVS alone (Usual Care (UC). The investigators will recruit 90 adults (30 per site) over the targeted recruitment period of approximately 6 months. The primary outcome of interest is the feasibility of the trial and acceptability of the AUDIO intervention. The investigators will also explore the impact of AUDIO on patients' ability to self-manage care (as well as other exploratory health-related outcomes and healthcare utilization) at regular intervals from enrollment (T1 = 1 week, T2 = 3 months) compared to baseline (T0 = pre-visit) and usual care. The investigators will recruit patients from consented clinicians at three sites: Dartmouth-Hitchcock Primary Care (D-H; Manchester, NH), Vanderbilt University Medical Center (VUMC; Nashville, TN), and University of Texas Medical Branch, (UTMB; Galveston, TX).

DETAILED DESCRIPTION:
Up to eighty percent of clinic visit information is forgotten by patients immediately post-visit. This is a significant barrier to self-management, especially in older adults with multimorbidity leading to poor health outcomes. After visit summaries (AVS) can improve recall, yet concerns exist about their layout, accuracy and low patient uptake. Patients and clinicians have begun audio recording clinic visits. When patients receive an audio recording of the visit, 71% listen and 68% share it with a caregiver, resulting in greater recall. Despite its growing use, to date, there is no research on the impact of recording and sharing clinic visits of patient self-management ability, health-related outcomes or healthcare utilization. The objective of this proposal is to conduct a multi-site pilot trial evaluating the feasibility and acceptability of routinely sharing audio recordings of clinic visits (AUDIO) in older adults (≥65 years) with diabetes and hypertension.

Conduct a multi-site, two-arm, parallel-group, patient-randomized, blocked, controlled, pilot trial with 3-month follow up, to determine the feasibility and acceptability of sharing audio recordings of clinic visits (AUDIO) on self-management in older adults with diabetes and hypertension, compared to the after visit written summary (AVS) alone (Usual Care). Investigators will determine:

1.1 Feasibility of a larger trial by meeting recruitment targets at each site (n=30 per site; total n=90) and determining the optimal strategy to achieve a high retention rate and adherence to the study protocol.

1.2 Acceptability by assessing the proportion of patients and clinicians who agree to take part in the project and the proportion of patients who listen to the recording.

1.3 Potential effectiveness by collecting data on the impact of audio recordings on self-management, health-related outcomes, healthcare utilization, and clinician behavior. Investigators hypothesize that compared to those receiving UC, patients randomized to also receive audio recordings (AUDIO) of clinic visits will report a greater self-management activation (Patient Activation Measure - Short Form) at 3 months. Investigators will also explore whether the effect of AUDIO on self-management activation compared to UC is greater for patients with low health literacy than those with high health literacy.

ELIGIBILITY:
Aim 1 Inclusion Criteria

* Age 65 years or older
* Diagnosed with diabetes mellitus (Type 1 or 2) and hypertension, and receiving medication for both
* Are patients of clinicians at the study clinic
* Have had one or more clinic visits in the previous seven months
* Plan on receiving care at the study clinic for the next six months

Exclusion Criteria

* Without the capacity to provide informed consent
* Diagnosis of dementia
* Diagnosis of schizophrenia and other psychotic disorders
* Current substance-abuse use disorder
* Diagnosis of an uncorrectable hearing or visual impairment, with no adjustments to support accessing the interventions or surveys
* Six item screener of cognitive function score 4 or less
* Living in a skilled nursing home or hospice
* Have audio-recorded a clinic visit for personal use within the past six months
* Do not have a personal email, do not have an email address shared with a family member or patient-identified caregiver, and/or are not willing to create an email account between the first contact from the study team and the initiation of online recording software registration

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Barr, PhD, Principal Investigator — Dartmouth College; Kerri L Cavanaugh, MD, Principal Investigator — Vanderbilit University Medical Center; Meredith C Masel, PhD, Principal Investigator — University Texas Medical Branch
Locations (3):
- United States (3):
  - Dartmouth-Hitchcock Manchester, Manchester, New Hampshire
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of results in peer-reviewed journals, access to the de-identified data for research purposes will be considered if a request is made by a qualified individual (i.e., a researcher from a research institute), IRB secured, and mutually agreed upon by the PIs. Any potential users of the data will sign an agreement that no attempt to reveal personal or private information may be made. The investigators will follow the Safe Harbour Methods outlined in the guidance regarding methods for de-identification of protected health information in accordance with the HIPAA Privacy Rule.
Supporting Information: Study Protocol
Time Frame: At the completion of data analysis
Access Criteria: Contact PI to request data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment began with study clinicians who were recruited beginning in August 2020. Patient participants were recruited from study clinicians at three academic medical center-affiliated primary care clinics between October 2020 and September 2021. Letters were sent to potentially eligible patients, and after a two-week opt-out period, study coordinators contact patients to determine the patient's interest in the project and eligibility.
Pre-assignment Details: Of 420 potential patients who received a mailed study invitation letter, we recruited 91: 120 patients were ineligible; 15 patients opted out; 122 declined during a screening call; 65 could not be reached and 7 could not take part for other reasons
Groups:
- AUDIO: Participant clinic visits will be audio recorded locally on a secure, HIPAA-compliant server. Patient access to recordings will be performed via a secure web-based platform.
  Additionally, participants will be offered the After Visit Summary (AVS) prior to clinic departure, per Usual Care (UC)
  Audio recording: The investigators will audio record the visits of patients in the intervention group. An RA will enter the exam room and begin the recording with the patient's permission. The patient and clinician can choose to stop or start the recording at any time. Once the visit is complete, the RA will enter the room, turn off the recording, and bring the patient to a private room where the RA will follow standardized instructions demonstrating how to access recordings. Patient access to recordings will be possible via a secure web-based platform. Patients will also receive reminders to listen to their recordings.
Period: Overall Study
Arm/Group | AUDIO | Usual Care
Started | 45 | 46
Completed | 44 | 45
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AUDIO | Usual Care | Total
Number analyzed (Participants) | 45 | 46 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.7 (5.8) | 73.7 (5.6) | 73.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 32 | 59
  Male | 18 | 14 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 39 | 43 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 37 | 38 | 75
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 45 | 46 | 91

OUTCOME MEASURES:

1. Primary Outcome: Participant Retention (Feasibility)
Description: The proportion of included participants completing the 3-month (T2) follow up assessment.
Time Frame: 3 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | AUDIO | Usual Care
Number analyzed (Participants) | 45 | 46
Participants | 44 | 45

2. Primary Outcome: Intervention Fidelity (Feasibility)
Description: The proportion of participants in the intervention arm that received the audio recording intervention with full adherence to a pre-defined protocol fidelity checklist. Any deviations will be documented.
Time Frame: 3 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | AUDIO
Number analyzed (Participants) | 45
Participants | 42

3. Primary Outcome: Feasibility of Intervention Measure (FIM)
Description: The FIM is a four-item patient-reported measure of intervention feasibility. Each item is scored from 1 (completely disagree) to 5 (completely agree), with a higher score indicating greater feasibility. We consider a score of ≥ 3 or higher to indicate the acceptable Feasibility of the intervention. We report the proportion of patients in the Intervention arm who scored ≥ 3.
Time Frame: 3 months from baseline
Population: Of 45 patients assigned to the Intervention arm, 42 completed the FIM survey. As such the overall number of participants analyzed for this outcome is 42.
Measure: Count of Participants; unit: Participants
Arm/Group | AUDIO
Number analyzed (Participants) | 42
Participants | 41

4. Primary Outcome: Participant Recruitment Rate (Acceptability)
Description: We considered our trial to be acceptable to patients if we could meet recruitment targets at each site of 30 patients. We also calculated our recruitment rate based on the number of potentially eligible patients contacted.
Time Frame: Baseline
Population: Of 420 potential patients who received a mailed study invitation letter, we recruited 91; 120 patients were ineligible; 15 patients opted out; 122 declined during a screening call; 65 could not be reached and 7 could not take part for other reasons (e.g., natural disaster, study staff COVID Quarantine). This resulted in 228 potentially eligible patients.
Measure: Count of Participants; unit: Participants
Groups:
- Potentially Eligible Patients: We calculated the recruitment rates based on the proportion of potentially eligible patients recruited.
Arm/Group | Potentially Eligible Patients
Number analyzed (Participants) | 228
Participants | 91

5. Primary Outcome: Intervention Use (Acceptability)
Description: The proportion of participants in the intervention arm that listen to the recordings received during the study period.
Time Frame: 3 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | AUDIO
Number analyzed (Participants) | 45
Participants | 40

6. Primary Outcome: Acceptability of Intervention Measure (AIM)
Description: The AIM is a four-item patient-reported measure of intervention acceptability. Each item is scored from 1 (completely disagree) to 5 (completely agree), with a higher score indicating greater acceptability. We consider a score of ≥ 3 or higher to indicate adequate acceptability of the intervention. We report the proportion of patients in the Intervention arm who scored ≥ 3.
Time Frame: 3 months from baseline
Population: Of 45 patients assigned to the Intervention arm, 42 completed the AIM survey. As such the overall number of participants analyzed for this outcome is 42.
Measure: Count of Participants; unit: Participants
Arm/Group | AUDIO
Number analyzed (Participants) | 42
Participants | 39

7. Other Pre Specified Outcome: Patient Activation Measure-Short Form (PAM-SF)
Description: The Patient Activation Measure-Short Form is a 13-item patient reported measure. Scores range from 0 (low activation) to 100 (high activation).
Time Frame: 3-Months from enrollment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Interpersonal Processes of Care Scale (IPC)
Description: Interpersonal Processes of Care Scale is an 18-item patient-reported measure assessing 7 sub-domains of interpersonal communication (Hurried communication; Elicited concerns, responded; Explained results, medications; Patient-centered decision making; Compassionate, respectful; Discrimination; Disrespectful office staff ). Direction of scoring: All scales are scored so that higher scores indicate higher frequency of the labeled interpersonal process. Thus, higher scores sometimes indicate better processes (e.g., decided together) and sometimes worse processes (e.g., lack of clarity). Calculating scores: All IPC items use an identical set of response options: 1='never'; 2='rarely'; 3='sometimes'; 4='usually'; 5='always.' Scale scores are calculated as the mean of non-missing responses to the corresponding items (i.e., item responses are averaged). Thus, scores have a possible range of 1-5 and can be calculated for an individual if at least one item per scale has a valid response.
Time Frame: 1-Week from baseline visit
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Patient Satisfaction Questionnaire-18 (PSQ-18)
Description: Patient Satisfaction Questionnaire-18 is a patient reported measure of satisfaction with seven dimensions: general satisfaction; technical quality; interpersonal manner; communication; financial aspects; time spent with doctor; accessibility and convenience. Responses are on a 5-point scale (Strongly agree - strongly disagree). Scores are averaged between 1 - 5; items 1,2,3,5,6,8,11,15,18 should be reversed scored i.e., 1 to 5, 2 to 4, 4 to 2, 5 to 1. Higher agreement reflects higher satisfaction with care.
Time Frame: Baseline,1-Week, and 3-Months from enrollment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Medical Outcomes Study General Adherence Measure
Description: The Medical Outcomes Study General Adherence measure, is a five-item patient reported measure of general treatment adherence.
Time Frame: 3-Months from enrollment
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Adherence to Refills and Medications (ARMS- 7)
Description: Adherence to Refills and Medications is a Seven-item patient reported measure of medication adherence.
Time Frame: 3-Months from enrollment
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Global PROMIS-10
Description: Global PROMIS (Patient-Reported Outcome Measurement Information System) is a 10-item patient reported measure with two domains: mental and physical health.
Time Frame: 3-Months from enrollment
Reporting Status: Not Posted

13. Other Pre Specified Outcome: EURO-QoL (EQ-5D)
Description: EURO-QOL is patient reported measure of quality of life (QOL) that can be calculated using responses to Global PROMIS.
Time Frame: Baseline,1-Week, and 3-Months from enrollment
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Primary Care Contact, ER Visits & Hospitalization
Description: Information on primary care contacts (phone calls, visits), ER visits & hospitalization will be collected via EMR. Baseline assessment will calculate primary care contacts, ER visits & hospitalization for each participant.
Time Frame: 3-Months from enrollment
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Quality of Diabetes and Hypertension Care
Description: Information on quality of diabetes and hypertension, including referrals to specialists and intensification of medication therapy, will be collected via EMR.
Time Frame: 3-Months from enrollment
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Patient Health Questionnaire (PHQ- 8)
Description: The eight-item depression scale PHQ-8 is a patient-reported multipurpose instrument to diagnose and measure the severity of depression. Scores range from 0 (no symptoms) - 24 (severe symptoms).
Time Frame: Baseline,1-Week, and 3-Months from enrollment
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Generalized Anxiety Disorder (GAD-7)
Description: The seven-item GAD-7 is a patient reported measure assessing severity of anxiety.
Time Frame: 3-Months from enrollment
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Comprehensive Diabetes Stigma Scale (CDSS-15)
Description: The comprehensive diabetes stigma scale (CDSS-15) is a validated 15-item assessment of diabetes-related stigma.
Time Frame: Baseline,1-Week, and 3-Months from enrollment
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Stigma Scale for Chronic Illness (SSCI-8)
Description: The Stigma Scale for Chronic Illness (SSCI-8) is validated, eight-item assessment of stigma related to chronic disease.
Time Frame: Baseline,1-Week, and 3-Months from enrollment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | AUDIO | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/45 | 1/46
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/46
Other Adverse Events (participants affected / at risk) | 0/45 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT04344301/Prot_SAP_ICF_000.pdf